CLINICAL TRIAL: NCT05492162
Title: An Intervention to Promote Health Students' Well-being : a Protocol of a Quasi-experimental Interventional Study in Le Havre
Brief Title: An Intervention to Promote Health Students' Well-being
Acronym: IFPDays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IFPDays
Record Dates: First submitted 2022-07-26; First posted 2022-08-08 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Healthy Lifestyle; Students Wellbeing
Keywords: health promotion; wellness program; health occupations students

STUDY DESIGN:
Intervention Model Description: before/after study using a quasi-experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- paramedic students (Other): para-experimental arm
  Interventions: Other: well-being promotion intervention

INTERVENTIONS:
Other: well-being promotion intervention — The intervention will be organized on both conferences and workshops.
  Four themes will be covered :
  * Well-being (Workshops)
  * Smoking prevention (Conference)
  * Balanced diet (Workshop)
  * Optimal organization for daily healthy living (Conference)

SUMMARY:
The lack of well-being observed among health students underscores the urgent need of implementing interventions designed to meet their specific need and improving their quality of life.

This study aims to evaluate a well-being promotion intervention among paramedic students.

This is a before/after study using a quasi-experimental design. This study aims to compare well-being, resilience, and self-esteem before and after the intervention.

Students' satisfaction will be assessed through a questionnaire.

DETAILED DESCRIPTION:
Health students' well-being is a big issue today. We need to increase the number of interventions designed to improve quality of life and well-being among this population of students.

The investigators aim to evaluate a well-being promotion intervention among paramedic students through a before/after study using a quasi-experimental design by comparing the scores of validated scales of well-being, resilience, and self-esteem of participating students before and after the intervention.

A satisfaction questionnaire will allow to assess the content and the organization of this intervention.

The first edition will be implemented in September 2022 in Le Havre. The questionnaires will be distributed before and eight months after the intervention.

The investigators will describe the study population, then they will compare the average scores.

The results of satisfaction questionnaire will allow to improve the intervention to best meet the needs of students.

The main benefit expected from this study is the improvement of paramedic students' well-being by adopting a healthy lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* paramedic students enrolled at IFP Mary Thieullent in september 2022

Exclusion Criteria:

* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Well-being | Month 1 and Month 8
  Change of average scores of Warwick-Edinburgh Mental Wellbeing Scale - 14 items Scores from 14 to 70: the higher score indicates a better wellbeing

SECONDARY OUTCOMES:
Resilience | Month 1 and Month 8
  Change of average scores of Connor-Davidson Resilience scale - 10 items Scores from 0 to 40: the higher score indicates a strong resilience
Self-esteem | Month 1 and Month 8
  Change of average scores of Rosenberg scale - 10 items Scores from 10 to 40 : the higher score indicates a better self-esteem
Students' Satisfaction | Month 1
  Satisfaction data will be analyzed to identify the strengths and the areas for improving the intervention (qualitative and qualitative analyses)

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier du Havre, Le Havre, France

IPD SHARING:
Plan to Share IPD: No